CLINICAL TRIAL: NCT04793997
Title: Covid-19 Primary Care Support With Microbiome Therapy.
Brief Title: Microbiome Therapy in Covid-19 Primary Care Support
Acronym: MiCel
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Based on feedback from our study participants on the taste, spray optimization is necessary
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Sarah Lebeer, Prof. dr.ir., Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B3002021000018
Record Dates: First submitted 2021-02-28; First posted 2021-03-11 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: SARS-CoV Infection; Corona Virus Infection
Keywords: lactobacilli; Probiotics; Throat spray
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verum Microbiome spray group (Active Comparator): Daily use of microbiome spray for two weeks
  Interventions: Biological: Microbiome spray
- Placebo spray group (Placebo Comparator): Daily use of placebo spray for two weeks
  Interventions: Biological: Placebo spray
- Household member group (No Intervention): No use of spray

INTERVENTIONS:
Biological: Microbiome spray — Throat spray containing 3 beneficial lactobacilli strains
  Arms: Verum Microbiome spray group
Biological: Placebo spray — Throat spray
  Arms: Placebo spray group

SUMMARY:
This double-blind, randomized, placebo-controlled study aims to investigate whether a throat spray containing probiotic bacteria (i.e. microbiome spray) can reduce the symptoms and complaints of the SARS-CoV-2 virus in patients with mild to moderate symptoms. In addition, the aim is to investigate whether the microbiome spray can prevent transmission of the SARS-CoV-2 virus to household members.

ELIGIBILITY:
Inclusion Criteria:

* Patients in primary care with a positive SARS-CoV-2 test based on PCR
* Instructed during screening and agreed not to use other probiotic nutritional supplements outside of the study during the study period
* Sign the consent form

Exclusion Criteria:

* Antibiotic use at baseline and during the study
* Vaccinated against SARS-CoV-2 at start of the study (both for index patients and household members that participate)
* Pregnant women
* History of use of probiotic supplements in the past two weeks
* Current diagnosis of cancer or immunosuppressive therapy within the past 6 months
* Acute and chronic infectious and inflammatory upper airway diseases (eg acute / chronic rhinosinusitis)
* Clinically significant bleeding disorder
* Any other medical condition that, in the principal investigator's opinion, warrants exclusion from the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in severity of COVID-19 infection symptoms after using microbiome spray | 3 weeks
  Change in severity of COVID-19 infection symptoms as assessed by a symptom score (min 0 - max 65) based on the presence and absence of fever and ten COVID-19 related symptoms and, if present, the four and five severity categories, respectively.

SECONDARY OUTCOMES:
Change in duration of COVID-19 infection symptoms after using microbiome spray | 3 weeks
  Change in duration of COVID-19 infection symptoms as assessed by a symptom score (min 0 - max 65) based on the presence and absence of fever and ten COVID-19 related symptoms and, if present, the four and five severity categories, respectively.
Change in absolute numbers of SARS-CoV-2 after using microbiome spray | 3 weeks
  Quantification via qPCR
Change in absolute numbers of specific bacterial pathogens after using microbiome spray | 3 weeks
  Quantification via qPCR
Change in microbiome of nose/throat region after using microbiome spray. | 3 weeks
Prevalence of antibodies against SARS-CoV-2 in the index patients' household members | 3 weeks
  The investigators will assess the prevalence of antibodies against SARS-CoV-2 in the index patients' household members based on the analysis of a capillary (fingerprick) blood sample stored on Whatman903 protein saver card
Prevalence of COVID-19 in the index patients' household members | 3 weeks
  The investigators will assess the prevalence of COVID-19 in the index patients' household members based on the presence of symptoms reported in a symptom diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Veronique Verhoeven, Antwerp, Belgium